CLINICAL TRIAL: NCT03749928
Title: OstiSense Biosensor in Bruxism Reduction - A Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0533276
Record Dates: First submitted 2018-11-12; First posted 2018-11-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Bruxism, Sleep
Keywords: night guard; biofeedback; biosensor
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- OstiSense biosensor - active (Experimental): Participants will wear the biofeedback tool for 1 week with biofeedback turned off. After checking, for 3 more weeks the biofeedback will stay turned off. At 4-week recall the biofeedback mechanism will be turned on. Subjects will be instructed how to use the vibration mechanism. Participants will wear the tool with biofeedback turned on during the night/sleep for 8 more weeks. They will be asked to return for a check after the first week with biosensor turned on (5-week recall). At the end of 8 weeks, participants will be invited for a final recall visit (12-week recall). At points a questionnaire will be provided, and feedback questions will be asked. All data about bruxism episodes will be collected from the smart device.
  Interventions: Device: OstiSense biosensor - active
- OstiSensor biosensor - not activated (Placebo Comparator): Participants in the control group will be treated, asked for feedback and receive questionnaires identical to the subjects in the active treatment group. The only difference will be that the biofeedback mechanism in the biofeedback night guard tool will always stay turned off. At the 1-week recall a check for any comfort issues will occur and accurate data recording will be confirmed. After three weeks the participant will be checked on, feedback will be requested and any wear issues will be identified, and the data recording function will be checked (4-week recall). At the end of additional 8 weeks participants will be invited for a final recall visit (12-week recall). A questionnaire will be provided, and feedback questions will be asked, data from the smart device about bruxism episodes will be collected.
  Interventions: Device: OstiSensor biosensor - not activated

INTERVENTIONS:
Device: OstiSense biosensor - active — The activated biofeedback back night guard will be used to reduce sleep bruxism
  Arms: OstiSense biosensor - active
Device: OstiSensor biosensor - not activated — A not-activated night guard will be used as control device
  Arms: OstiSensor biosensor - not activated

SUMMARY:
The overall objective of the clinical studies with the OstiSense biosensor tool will be to evaluate whether the use of the OstiSense biosensor tool significantly reduces the number of sleep bruxism events per night as well as the duration of those events for patients with bruxism.The product under investigation is the OstiSense biosensor with biofeedback for bruxism therapy. The sensor is integrated in a night-guard like device and registers the pressure created during a bruxism episode. If a predetermined pressure threshold is exceeded, the integrated vibration tool will be activated, and the vibrations will/should remind the wearer to stop clenching his jaws and relax his facial muscles. Due to this feedback, the number of bruxism episodes as well as clenching time per episode should be reduced. The sensor also identifies the time of grinding and the sleep stage of the patient.

DETAILED DESCRIPTION:
Pilot Study:

30 subjects will be recruited for this pilot study. An oral exam will be performed to check for gingiva and tooth conditions as well as fulfilling inclusion and exclusion criteria as described below. Subjects will be randomly assigned to an active treatment or a control group. OstiSense biosensor feed back tool (night guards) will be delivered to the participant. First patient impressions about wearing comfort will be evaluated, chair side. Then the investigators will test the efficiency of the OstiSense biosensor feedback tool in reduction of numbers of bruxism episodes and reduction of the duration of bruxism episodes (primary outcome). These data will be collected also in order to achieve information for a sample size calculation for a larger subsequent clinical trial. The investigators will collect information about self-reported (or reported by sleeping partners in SB) reduced frequency of bruxism episodes. In addition, self-reported reduction in pain (facial pain, myofascial headache) (secondary outcome) is of interest. Visual pain scales and pain questionnaires will be used as validated instruments for subjective pain assessment.

Active Treatment Group:

Participants will be instructed to wear the biofeedback tool during the night/sleep. They will wear the biofeedback tool for 1 week with biofeedback turned off to record baseline activity. At the 1-week recall, the investigators will check for any comfort issues and will confirm accurate data recording. For 3 more weeks the biofeedback will stay turned off to collect further baseline data.

At the next recall (4-week recall) participants will be interviewed about any wear issues and will be asked to fill out the same questionnaire as used in phase 1 of the pilot study. The biofeedback mechanism will then be turned on (battery insertion). During this meeting subjects will be instructed to test the vibration mechanism by increasing their bite force until vibration occurs, and then to relax their muscles so that vibration stops. Subjects will be asked to repeat this procedure several times to get familiar with the active device and also to learn to relax their muscles when the feedback occurs during night bruxism..

Participants will wear the tool with biofeedback turned on during the night/sleep for 8 more weeks. They will be asked to return for a check after the first week (5-week recall) of the 8 weeks to identify any wear issues while the tool is turned on, and for checking the data recording function. At the end of 8 weeks, participants will be invited for a final recall visit 12-week recall). The same questionnaire will be provided, and feedback questions will be asked. All data about bruxism episodes will be collected from the smart device.

Control Group:

Participants in the control group will be treated, asked for feedback and receive questionnaires identical to the subjects in the active treatment group. The only difference will be that the biofeedback mechanism in the biofeedback night guard tool will always stay turned off. At the 1-week recall the investigators will check for any comfort issues and will confirm accurate data recording. After three weeks the investigators will again check on the participant, will identify any wear issues, ask for feedback and will check the data recording function (4-week recall). At the end of additional 8 weeks participants will be invited for a final recall visit (12-week recall). The questionnaire will be provided, and feedback questions will be asked. Data from the smart device about bruxism episodes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years, in good general health
* the occlusion is stable with at least 8 lower teeth (including several lower front teeth)
* willing to comply with all study procedures and protocols
* must be able to read and understand English
* have an understanding of the study
* able to provide written informed consent in English
* willing to sign the "Authorization for Release of Personal Health Information and Use of Personally Unidentified Study Data for Research" form; data will only be used for research.

Exclusion Criteria:

* having acute temporo mandibular joint pain or a history of acute temporo mandibular joint pain
* having used a biofeedback tool for bruxism reduction before
* subjects not having a smart phone device
* subjects not willing to use their smart phone device for data collection related to their bruxism
* heavily crowed lower teeth (difficult to integrate a night guard)
* wearing complete dentures
* show evidence of extremely poor oral hygiene
* subjects at extreme high caries risk
* subjects with pacemakers
* subjects suffering from systemic diseases, significant past or medical history with conditions that may affect oral health or oral flora (i.e. diabetes, HIV, heart conditions that require antibiotic prophylaxis),
* taking medications that may affect the oral flora or salivary flow (e.g. antibiotic use in the past three months, drugs associated with dry mouth / xerostomia [extreme high caries risk])
* other conditions that may decrease the likelihood of adhering to study protocol
* subjects who will leave the area and are unable to complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of bruxism episodes | 8 weeks
  Evaluating how efficient the OstiSense biosensor tool is in changing the number of bruxism episodes
Change in duration of bruxism episodes | 8 weeks
  Evaluating how efficient the OstiSense biosensor tool is in changing the duration of bruxism episodes

SECONDARY OUTCOMES:
Self-reported change in frequency of bruxism episodes | 8 weeks
  Self-reported (or reported by sleeping partners in SB) change in frequency of bruxism episodes
Self-reported change in pain - change in pain level marked on a visual pain scale | 8 weeks
  Self-reported change in pain (facial pain, myofascial headache) assessed using a visual pain scale with 6 different pain levels indicated by 6 different smileys (from happy smiling to crying) and a pain severity scale from 0 to 10, which includes the smiley faces, with 0 as no pain, 1-2 slight pain, 3-4 mild, 5-6 moderate, 7-8 severe and 9-10 horrible pain
Self-reported change in pain - change in yes/no answers on a pain questionnaire | 8 weeks
  Self-reported change in pain (facial pain, myofascial headache) using a pain questionnaires requiring yes and no answers to questions

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rechmann, DMD, PhD, Principal Investigator — UCSF School of Dentistry
Locations (1):
- UCSF School of Dentistry - Dental Offices in Bay Area, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, de Leeuw R, Manfredini D, Svensson P, Winocur E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013 Jan;40(1):2-4. doi: 10.1111/joor.12011. Epub 2012 Nov 4. PMID 23121262
- [Background] Carra MC, Huynh N, Lavigne G. Sleep bruxism: a comprehensive overview for the dental clinician interested in sleep medicine. Dent Clin North Am. 2012 Apr;56(2):387-413. doi: 10.1016/j.cden.2012.01.003. PMID 22480810
- [Background] Svensson P, Jadidi F, Arima T, Baad-Hansen L, Sessle BJ. Relationships between craniofacial pain and bruxism. J Oral Rehabil. 2008 Jul;35(7):524-47. doi: 10.1111/j.1365-2842.2008.01852.x. PMID 18557918
- [Background] de la Hoz-Aizpurua JL, Diaz-Alonso E, LaTouche-Arbizu R, Mesa-Jimenez J. Sleep bruxism. Conceptual review and update. Med Oral Patol Oral Cir Bucal. 2011 Mar 1;16(2):e231-8. doi: 10.4317/medoral.16.e231. PMID 21196839
- [Background] Koyano K, Tsukiyama Y, Ichiki R, Kuwata T. Assessment of bruxism in the clinic. J Oral Rehabil. 2008 Jul;35(7):495-508. doi: 10.1111/j.1365-2842.2008.01880.x. PMID 18557916
- [Background] Ilovar S, Zolger D, Castrillon E, Car J, Huckvale K. Biofeedback for treatment of awake and sleep bruxism in adults: systematic review protocol. Syst Rev. 2014 May 2;3:42. doi: 10.1186/2046-4053-3-42. PMID 24886985
- [Background] Lavigne GJ, Khoury S, Abe S, Yamaguchi T, Raphael K. Bruxism physiology and pathology: an overview for clinicians. J Oral Rehabil. 2008 Jul;35(7):476-94. doi: 10.1111/j.1365-2842.2008.01881.x. PMID 18557915
- [Background] Bowley JF, Stockstill JW, Pierce CJ. Reliability and validity of instrumentation used to record nocturnal clenching and/or grinding. J Orofac Pain. 1993 Fall;7(4):378-85. PMID 8118441
- [Background] Rivera-Morales WC, McCall WD Jr. Reliability of a portable electromyographic unit to measure bruxism. J Prosthet Dent. 1995 Feb;73(2):184-9. doi: 10.1016/s0022-3913(05)80160-x. PMID 7722935
- [Background] Hublin C, Kaprio J, Partinen M, Koskenvuo M. Sleep bruxism based on self-report in a nationwide twin cohort. J Sleep Res. 1998 Mar;7(1):61-7. doi: 10.1046/j.1365-2869.1998.00091.x. PMID 9613429
- [Background] Molina OF, dos Santos J Jr, Nelson SJ, Grossman E. Prevalence of modalities of headaches and bruxism among patients with craniomandibular disorder. Cranio. 1997 Oct;15(4):314-25. doi: 10.1080/08869634.1997.11746026. PMID 9481994
- [Background] Gavish A, Halachmi M, Winocur E, Gazit E. Oral habits and their association with signs and symptoms of temporomandibular disorders in adolescent girls. J Oral Rehabil. 2000 Jan;27(1):22-32. doi: 10.1046/j.1365-2842.2000.00484.x. PMID 10632840
- [Background] Lobbezoo F, van der Zaag J, van Selms MK, Hamburger HL, Naeije M. Principles for the management of bruxism. J Oral Rehabil. 2008 Jul;35(7):509-23. doi: 10.1111/j.1365-2842.2008.01853.x. PMID 18557917
- [Background] Jagger R. The effectiveness of occlusal splints for sleep bruxism. Evid Based Dent. 2008;9(1):23. doi: 10.1038/sj.ebd.6400569. PMID 18364692
- [Background] Macedo CR, Silva AB, Machado MA, Saconato H, Prado GF. Occlusal splints for treating sleep bruxism (tooth grinding). Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005514. doi: 10.1002/14651858.CD005514.pub2. PMID 17943862
- [Background] Macedo CR, Macedo EC, Torloni MR, Silva AB, Prado GF. Pharmacotherapy for sleep bruxism. Cochrane Database Syst Rev. 2014 Oct 23;2014(10):CD005578. doi: 10.1002/14651858.CD005578.pub2. PMID 25338726
- [Background] Klasser GD, Greene CS, Lavigne GJ. Oral appliances and the management of sleep bruxism in adults: a century of clinical applications and search for mechanisms. Int J Prosthodont. 2010 Sep-Oct;23(5):453-62. PMID 20859563
- [Background] Rosar JV, Barbosa TS, Dias IOV, Kobayashi FY, Costa YM, Gaviao MBD, Bonjardim LR, Castelo PM. Effect of interocclusal appliance on bite force, sleep quality, salivary cortisol levels and signs and symptoms of temporomandibular dysfunction in adults with sleep bruxism. Arch Oral Biol. 2017 Oct;82:62-70. doi: 10.1016/j.archoralbio.2017.05.018. Epub 2017 May 27. PMID 28601734
- [Background] Rugh JD, Johnson RW. Temporal analysis of nocturnal bruxism during EMG feedback. J Periodontol. 1981 May;52(5):263-5. doi: 10.1902/jop.1981.52.5.263. PMID 6941011
- [Background] Cassisi JE, McGlynn FD, Belles DR. EMG-activated feedback alarms for the treatment of nocturnal bruxism: current status and future directions. Biofeedback Self Regul. 1987 Mar;12(1):13-30. doi: 10.1007/BF01000075. PMID 3311171
- [Background] Gu W, Yang J, Zhang F, Yin X, Wei X, Wang C. Efficacy of biofeedback therapy via a mini wireless device on sleep bruxism contrasted with occlusal splint: a pilot study. J Biomed Res. 2015 Apr;29(2):160-8. doi: 10.7555/JBR.28.20130145. Epub 2014 Nov 18. PMID 25859272
- [Background] Foster PS. Use of the Calmset 3 biofeedback/relaxation system in the assessment and treatment of chronic nocturnal bruxism. Appl Psychophysiol Biofeedback. 2004 Jun;29(2):141-7. doi: 10.1023/b:apbi.0000026640.54839.83. PMID 15208977
- [Background] Wang LF, Long H, Deng M, Xu H, Fang J, Fan Y, Bai D, Han XL. Biofeedback treatment for sleep bruxism: a systematic review. Sleep Breath. 2014 May;18(2):235-42. doi: 10.1007/s11325-013-0871-y. Epub 2013 Jun 12. PMID 23756884